CLINICAL TRIAL: NCT02683629
Title: A Phase IIb, Randomised, Double-blind, Placebo-controlled, Dose-range Investigation of the Safety and Efficacy of NTCELL® [Immunoprotected (Alginate-Encapsulated) Porcine Choroid Plexus Cells for Xenotransplantation] in Patients With Parkinson's Disease
Brief Title: Investigation of the Safety and Efficacy of NTCELL® [Immunoprotected (Alginate-Encapsulated) Porcine Choroid Plexus Cells for Xenotransplantation] in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Living Cell Technologies (Industry)
Collaborators: Statistecol Consultants Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCT/PD-015
Record Dates: First submitted 2016-02-08; First posted 2016-02-17 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Xenotransplantation; choroid plexus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NTCELL (Experimental): NTCELL Implantation
  Interventions: Biological: NTCELL Implantation
- Sham Surgery (Sham Comparator): Sham Surgery
  Interventions: Other: Sham Surgery

INTERVENTIONS:
Biological: NTCELL Implantation — NTCELL Implantation
  Arms: NTCELL
Other: Sham Surgery — Sham Surgery
  Arms: Sham Surgery

SUMMARY:
To assess the safety of xenotransplantation of NTCELL [immunoprotected (alginate-encapsulated) choroid plexus cells] in patients with Parkinson's disease, assessed over the duration of the study, by monitoring the occurrence of adverse events and serious adverse events, including clinical and laboratory evidence of xenogeneic infection in transplant recipients and their partners/close contacts. Subsequent safety follow-up will include lifelong monitoring for clinical and laboratory evidence of xenogeneic infection.

To assess the efficacy of xenotransplantation of NTCELL [immunoprotected (alginate-encapsulated) choroid plexus cells] in patients with Parkinson's disease. This will be quantified by testing the secondary endpoints of the trial as described below (see Endpoints/Outcome Measures).

DETAILED DESCRIPTION:
Parkinson's disease is characterized by widespread neural degeneration, particularly in the substantia nigra and its projections to the basal ganglia. Current therapy for Parkinson's disease is purely symptomatic. There is a pressing need for a treatment that reverses or slows the degeneration of the nigrostriatal pathway.

Numerous transplant-based therapies have attempted to support, repair or replace the degenerating nigrostriatal neurons. These have included the transplantation of foetal and other neuronal stem cells, gene transfers, and the implantation of devices releasing neural growth factors. All these have been shown to have some effectiveness in animal models, but have been generally disappointing in human studies.

Intracranial choroid plexus cell transplantation has the potential to deliver biological neural agents for the treatment of Parkinson's disease which cannot be achieved by conventional treatment. The overall aim of delivering neural proteins and compounds over many months to the basal ganglia of the brain is to enhance neural repair currently not possible with antiparkinsonian medication or deep brain stimulation (DBS).

As animal-derived tissues have to be protected from immune rejection when transplanted into humans, transplants are usually accompanied by immunosuppressive therapy. However, porcine choroid plexus cells are preferably implanted without the use of immunosuppressive drugs which cause significant morbidity. To protect them from immune rejection, the cells can be encapsulated in alginate microcapsules which permit the inward passage of nutrients and the outward passage of biologic neural proteins and compounds normally secreted by choroid plexus cells. Alginate-encapsulated porcine choroid plexus cells implanted into the brain without immunosuppressive drugs have survived rejection for many months in animal studies.

NTCELL comprises neonatal porcine choroid plexus cells encapsulated in alginate microcapsules.

The bilateral dose that will be administered to the 18 patients (initially 3 groups of 6 patients, randomised 4:2 NTCELL:sham surgery) enrolled in this trial will be up to a total of twice the human equivalent dose administered unilaterally in LCT's non-human primate study. Thus up to 240 NTCELL microcapsules (± 5%) administered on each side of the brain.

If there are no significant safety issues after implantation of the first group of patients, the second group of patients will then be scheduled to receive implants of NTCELL.

If there are no significant safety issues after implantation of the second group of patients, the third group of patients will then be scheduled to receive implants of NTCELL.

This study will adopt an adaptive design in respect to the choice of dose of NTCELL for the fourth group of patients (those patients who originally received sham surgery in Groups 1-3). Following unblinding of the study after Groups 1-3 have reached 26-week follow-up, an interim analysis, for safety and efficacy, will be undertaken.

If there are no significant safety issues, the last group of patients, Group 4, (who originally received sham surgery) will be scheduled to receive NTCELL implants. The dose of NTCELL given will be determined by the DSMB following a proposal from the Principal Investigator, based on the results of the interim analysis.

Parkinson's disease patients will be followed up for 26 weeks after receiving either an implantation of NTCELL or sham surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (males or females) in the age range 40 to 65 years
2. Diagnosis of Parkinson's disease (minimum duration of 5 years) in accordance with the London Brain Bank criteria
3. Patients diagnosed with idiopathic Parkinson's disease
4. Optimum medication for Parkinson's disease
5. Expected to meet the criteria for DBS in the future, in the opinion of the Investigator
6. If female, no childbearing capability (those who are more than 2 years post-menopausal or have undergone voluntary sterilisation can be considered for enrolment)
7. Provision of written informed consent. Patients will be required to agree to comply with all tests and visits specified in the protocol, and they (and their partners/close contacts) will also be required to consent to long-term microbiological monitoring, which is an integral part of the study

Exclusion Criteria:

1. Any history of central nervous system infection
2. Significant dementia as determined by neuropsychiatric assessment
3. Focal neurological defects
4. Evidence of significant ongoing medical or psychiatric disorders
5. Secondary parkinsonism
6. Severe autonomic symptoms
7. Atypical Parkinson's disease
8. History of substance abuse
9. Body mass index (BMI) ≥ 30 kg/m2 or ≤ 20 kg/m2
10. Serious comorbid conditions that, in the opinion of the Investigator, are likely to affect participation in the study, including:

    1. Previous coronary heart disease manifesting as non-ST elevation myocardial infarction (NSTEMI), Q-wave infarction or unstable angina; coronary artery bypass graft (CABG); or percutaneous angioplasty
    2. Previous cerebrovascular disease manifesting as transient ischaemic attacks (TIAs) or stroke
    3. Peripheral vascular disease with foot ulcer and/or previous amputation
    4. History of New York Heart Association (NYHA) class II, III or IV congestive heart failure (CHF) and/or chronic atrial fibrillation
    5. Chronic obstructive pulmonary disease (COPD) or asthma with previous hospitalisation for decompensation; a requirement for mechanical ventilation at any stage; or long-term treatment with oral corticosteroids
    6. Liver disease with abnormal liver function tests defined as serum bilirubin ≥ 20 µmol/L, and/or ALT ≥ 100 U/L, and/or GGT ≥ 100 U/L, and/or albumin < 35 g/L
    7. Haematological disorders, including haemoglobin ≤ 110 g/L or platelet count < 80 x 109/L
    8. Kidney disease, defined as serum creatinine > 130 μmol/L in men and > 110 μmol/L in women and/or haematuria and/or active urinary sediment or casts
    9. Peptic ulcer disease and/or history of previous gastrointestinal bleeding
    10. Malignancy other than basal cell carcinoma
    11. History of epilepsy
    12. Untreated hypothyroidism
    13. Known adrenal insufficiency
11. Previous brain surgery for Parkinson's disease
12. Poor candidate for any surgery
13. HIV antibody and/or risk factors for HIV infection
14. Positive hepatitis C antibody, positive hepatitis B surface antigen, and hepatitis B core antibody
15. Current administration of immunosuppressive medications (e.g. cyclosporin, tacrolimus, sirolimus, mycophenolate mofetil, muromonab-CD3, daclizumab, basiliximab, antithymocyte globulin, interferons) for other disease conditions
16. Any other condition that, in the opinion of the Investigator, may interfere with adherence to the study protocol

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
The safety of xenotransplantation of NTCELL as measured by the incidence of adverse events related to treatment | up to 26 weeks
  Adverse events can result from, for example, abnormal clinical laboratory tests (including xenogeneic viral analysis), abnormal physical examination findings, any abnormal findings following review by an infectious disease physician. These multiple assessments result in the one outcome measure which is the incidence of treatment emergent adverse events

SECONDARY OUTCOMES:
Change in total Unified Parkinson's Disease Rating Scale (UPDRS in the 'off' and 'on' state) over 26 weeks post-intervention compared with baseline | Baseline and 26 weeks
Change in Unified Parkinson's Disease Rating Scale (UPDRS Part III in the 'on' state) over 26 weeks post-intervention compared with baseline | Baseline and 26 weeks
Change in Quality of life as assessed by Parkinson's Disease Questionnaire (PDQ-39) over 26 weeks post-intervention compared with baseline | Baseline and 26 weeks
Change in L-dopa dosage over 26 weeks post-intervention compared with baseline | Baseline and 26 weeks
Change in scores measured by the Unified Dyskinesia Rating Scale (UDysRS Parts I, II, III, IV - Parts III and IV will be performed in the 'off' and 'on' state) over 26 weeks post-intervention compared with baseline | Baseline and 26 weeks
Change in scores measured by the modified walking test in accordance with the CAPSIT-PD protocol (Defer et al. 1999) over 26 weeks post-intervention compared with baseline | Baseline and 26 weeks
Change in Modified Hoehn and Yahr stage over 26 weeks post-intervention compared with baseline | Baseline and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry Snow, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
International conference presentations, press releases, International journal publications